CLINICAL TRIAL: NCT07177274
Title: Evaluation of Skin Stiffness Changes in Wounds Before and After Low-Level Laser Therapy Using 660 nm Laser: A Comparative Analysis With OCT and MyotonPRO
Brief Title: Evaluation of Skin Stiffness Changes in Wounds Before and After Low-Level Laser Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NSTC 114-2923-E-468-001-MY3
Record Dates: First submitted 2025-09-10; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Wound - in Medical Care
Keywords: Stiffness; Wound; Skin; Low-Level Laser Therapy
MeSH Terms: conditions — Wounds and Injuries | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skin status (normal, wound, after treatment) (Active Comparator): Using 660 nm LLLT efficacy on the wound, separated categories into the upper limb and lower limb.
  Interventions: Radiation: Low Level Laser Therapy
- Skin location (upper limb, lower limb) (Active Comparator): Using 660 nm LLLT efficacy on the wound, separated categories into the upper limb and lower limb.
  Interventions: Radiation: Low Level Laser Therapy

INTERVENTIONS:
Radiation: Low Level Laser Therapy — Collecting wound stiffness data using the OCT-air-jet and Myoton Pro before and after the LLLT treatment using the device's indentation system. Then the intervention is applying LLLT to the wound for 3 min. The LLLT utilized the Red Dot Laser Diode Module Class IIIA.
  Other Names: 660 nm LLLT

SUMMARY:
Chronic wounds and impaired healing remain a major clinical challenge, particularly in patients with diabetes, vascular disease, or age-related skin fragility. Low-level laser therapy (LLLT) at 660 nm has been reported to enhance tissue repair, reduce inflammation, and promote angiogenesis. However, the biomechanical properties of wound tissue following LLLT remain poorly understood.

Optical Coherence Tomography (OCT) provides a non-invasive, high-resolution method to assess skin microstructure and elasticity, while the MyotonPRO offers quantitative stiffness measurements at the tissue surface. Combining these two complementary modalities may provide a more comprehensive assessment of wound healing progression and treatment response.

This study aims to evaluate changes in wound stiffness before and after 660 nm LLLT and to compare them against contralateral normal skin, thereby providing objective insight into the biomechanical efficacy of laser treatment.

ELIGIBILITY:
Inclusion Criteria:

* presented chronic and burn wounds lasting more than four weeks.
* had partial-thickness burn wounds.

Exclusion Criteria:

* current smokers.
* wounds that were fresh and still bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
To evaluate changes in skin stiffness of wound tissue before and after LLLT using OCT and MyotonPRO. | 1 year

SECONDARY OUTCOMES:
To compare wound skin stiffness with contralateral normal skin. | 1 year
  To assess differences in stiffness response between upper-body and lower-body wound sites.
  To determine the correlation between OCT and MyotonPRO stiffness measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Asia University, Taichung, Wufeng, Taiwan

IPD SHARING:
Plan to Share IPD: No